CLINICAL TRIAL: NCT00214201
Title: Campath-1H Induction to Allow Discontinuation of Calcineurin Inhibitors After Renal Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2003-125
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2012-09-12 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-09

CONDITIONS: Primary Renal Transplant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (No Intervention): Standard of Care CNI immunosuppression
- 2 (Experimental): Calcineurin inhibitor withdrawal
  Interventions: Drug: Calcineurin inhibitor withdrawal

INTERVENTIONS:
Drug: Calcineurin inhibitor withdrawal — stopping tacrolimus or cyclosporine in subjects who received Campath-1H induction therapy
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether Campath-1H induction therapy and the associated lymphocyte depletion will permit long-term, rejection free renal allograft function in the absence of maintenance calcineurin inhibitor (CI) therapy.

ELIGIBILITY:
Inclusion Criteria:

* received a renal transplant, induction with Campath-1H, and at least 2 months of calcineurin inhibitor therapy, CellCept, and prednisone.

Exclusion Criteria:

* Recipients of HLA-identical living-donor renal transplants;
* PRA value >20% within 30 days of transplant;
* GFR <40ml/min;
* multi-organ transplant;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2003-05; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Knechtle, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- CNI Control Post Campath 1H: Standard of Care CNI immunosuppression
- CNI Withdrawal Post Campath 1H: Calcineurin inhibitor withdrawal
  Calcineurin inhibitor withdrawal : stopping tacrolimus or cyclosporine in subjects who received Campath-1H induction therapy
Period: Overall Study
Arm/Group | CNI Control Post Campath 1H | CNI Withdrawal Post Campath 1H
Started | 20 | 20
Completed | 18 | 18
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Death | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CNI Control Post Campath 1H | CNI Withdrawal Post Campath 1H | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 17 | 33
  >=65 years | 4 | 3 | 7
Age Continuous [Mean (Standard Deviation); unit: years] | 54.1 (9.2) | 55.3 (9.4) | 54.7 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 17 | 15 | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Biopsy Proven Rejection
Time Frame: 3 years
Measure: Number; unit: participants
Groups:
- CNI Withdrawal Post Campath 1H: Calcineurin inhibitor withdrawal : stopping tacrolimus or cyclosporine in subjects who received Campath-1H induction therapy
Arm/Group | CNI Control Post Campath 1H | CNI Withdrawal Post Campath 1H
Number analyzed (Participants) | 20 | 20
participants | 2 | 7

2. Secondary Outcome: Serum Creatinine at 36 Months (End of Study)
Time Frame: 36 months +/- 60 days
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | CNI Control Post Campath 1H | CNI Withdrawal Post Campath 1H
Number analyzed (Participants) | 18 | 18
mg/dl | 1.49 (.44) | 1.37 (.35)

3. Other Pre Specified Outcome: WBC
Description: White Blood Cell count
Time Frame: 36 months +/- 60 days
Measure: Mean (Standard Deviation); unit: K/ul
Arm/Group | CNI Control Post Campath 1H | CNI Withdrawal Post Campath 1H
Number analyzed (Participants) | 18 | 18
K/ul | 7.10 (1.69) | 7.68 (2.05)

ADVERSE EVENTS:
Arm/Group | CNI Control Post Campath 1H | CNI Withdrawal Post Campath 1H
Serious Adverse Events (participants affected / at risk) | 11/20 | 8/20
Other Adverse Events (participants affected / at risk) | 10/20 | 11/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CNI Control Post Campath 1H (N=20) | CNI Withdrawal Post Campath 1H (N=20)
Atrial Fibrillaiton (Cardiac disorders) | 0 (0) | 1 (1)
encephalitis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Vascular disorders) | 0 (0) | 1 (3)
kidney transplant rejection (Immune system disorders) | 1 (1) | 2 (3)
back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — unknown etiology reuired hospitalization
hydronephrosis (Renal and urinary disorders) | 1 (1) | 3 (3)
cytomegalovirus (Infections and infestations) | 2 (2) | 2 (2) — required hospitalization
urinary tract infection (Renal and urinary disorders) | 1 (1) | 1 (1) — required hospitalization
thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
thryoidectomy (Surgical and medical procedures) | 0 (0) | 1 (1) — secondary to thyroid cancer
campylobacteremia (Infections and infestations) | 0 (0) | 1 (1)
hernia repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Idiopathic thrombocytopenic purpura (ITP), (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
congestive heart failure (Cardiac disorders) | 1 (1) | 0 (0)
Camplobacter gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
gastritis (viral) (Gastrointestinal disorders) | 1 (1) | 0 (0)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Coronary artery bypass grafting (CABG) (Surgical and medical procedures) | 1 (1) | 0 (0)
Varicella Zoster (Infections and infestations) | 1 (1) | 0 (0)
Cryptococcal Meningitis (Infections and infestations) | 1 (1) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CNI Control Post Campath 1H (N=20) | CNI Withdrawal Post Campath 1H (N=20)
Constipation (Gastrointestinal disorders) | 1 (2) | 0 (0)
urinary tract infection (Renal and urinary disorders) | 1 (1) | 3 (5)
Dental Abcess (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
BK Polyoma viuria (Infections and infestations) | 3 (3) | 2 (2)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Cytomegalovirus (Infections and infestations) | 1 (1) | 2 (2)
Upper Respiratory Tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Herpes Zoster (Infections and infestations) | 4 (4) | 1 (1)
E. Coli Urinary Tract Infection (Infections and infestations) | 2 (2) | 1 (1)
Klebsiella pneumoniae Urinary Tract infection (Infections and infestations) | 0 (0) | 1 (1)
Acinetobacter Baumannii Urinary Tract infection (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal Urinary Tract infection (Infections and infestations) | 0 (0) | 1 (1)
Iritis, left eye (Eye disorders) | 1 (1) | 0 (0)
CMV retinitis (Infections and infestations) | 1 (1) | 0 (0)
Epstein Barr Virus (Infections and infestations) | 1 (1) | 0 (0)
Boil (groin) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes